CLINICAL TRIAL: NCT04628702
Title: Playful Multimodal Intervention, Monitoring and Decision Support for Activation of People With Alzheimer's Dementia
Acronym: M-AAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Joanneum Research Forschungsgesellschaft mbH (Other); AustriaN Red Cross (OeRK) (Unknown); health system intelligence (HS & I) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FFG-Benefit 875345
Record Dates: First submitted 2020-10-28; First posted 2020-11-13 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; tablet-based multimodal training; longitudinal; efficacy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: two groups: interventional group with 1.5 years tablet training and a control group; both groups receive pre-post neurological, neuropsychological examination, MRI and blood sampling at study inclusion and 1.5 years later.
Who Masked: Investigator
Masking Description: Neurologist and neuropsychologist are not informed about intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): receives tablet-training
  Interventions: Behavioral: tablet training
- Control group (No Intervention): no training

INTERVENTIONS:
Behavioral: tablet training — 1.5 year training period
  Arms: Intervention group

SUMMARY:
The worldwide prevalence of dementia is increasing. Pharmaceutical therapies, at the best, slow the degenerative process, observable in Alzheimer's disease (AD). Additional approaches are therefore urgently needed to maintain the patient's independence and the abilities to execute activities of daily living to reduce the patient specific, familial and economic burden. Multimodal tablet-based training might be a potential linchpin in this quest. The primary aim of this study therefore is, to examine the efficacy of the tablet-based training program "Multimodal Activation" (MMA) in mild AD patients.

In a randomized controlled trial the investigators aim to include 220 mild AD patients, of which 110 are randomly assigned to the training group receiving guided tablet-based training for 1.5 years, and 110 to the control group. The multimodal intervention, as implemented in the training, includes physical, cognitive and social components. Efficacy of the training will be determined by means of between group pre-post comparison in quantitative neuropsychological and qualitative tests, MRI biomarker and blood biomarker.

DETAILED DESCRIPTION:
Background. The prevalence of Alzheimer's disease is increasing due to an aging society. Parallel, care and nursing needs and costs rise with disease progression. Promoting and stimulating patients to maintain patients abilities and the independent life is therefore essential to prolong the time at home and reduce direct and indirect costs. Computer-based technologies, such as tablet-based trainings, might have the potential to support the patient itself and the caregiver by reducing the (nursing) care-dependency and stabilizing or slowing the disease progression. Prior studies revealed that patients suffering from dementia in general desire technologies supporting cognitive abilities, communication skills, social integration and activities of daily living (e.g. mobility) (Lauriks et al .2007, Wand et al., 2016). Moreover, a multimodal approach has been demonstrated to be superior compared to unimodal approaches, aiming to foster only one domain or aspect. In this study, a multimodal tablet-based training, focusing on cognitive, psychological, physical and aspects of activities of daily living, for patients suffering from mild Alzheimer's disease was implemented.

The primary aim of this study is to examine the efficacy of the multi-domain approach which as implemented in the tablet-based training in mild AD patients. Secondary aims are to measures structural and functional cerebral changes, quality of life, mobility, motivation, life-style factors, stress, care-dependency, (instrumental) activities of daily living, changes in medical treatments, problems in behavior, burden due to nursing, activity level, arm strength, depressive symptoms and the usability of the data raised for the development of a decision support system.

Methods. This study is implemented as a randomized controlled trial with embedded design. Two-hundred twenty subjects with mild AD (dementia diagnoses according to NINCDS-ADRDA criteria) and the primary caregiver will be included in the study. One hundred ten subjects will receive a guided tablet-training for 1.5 years. One hundred ten subjects are in the control group, receiving "normal" medical treatment and support. Additionally, five nursing persons and 5 M.A.S. (Morbus Alzheimer syndrome) trainers conduct single and group trainings. All subjects and the caregivers will be tested and interviewed, respectively, at study entry, at six, twelve and eighteen months. The study team consist of Joanneum Research (JR), the Sozialverein Deutschlandsberg (SVDL), the Austrian Red Cross (ÖRK), and the Medical University of Graz, Department of Neurology and the Institute of Nursing Science as well as Health System & Intelligence (HS&I).

Recruiting. The recruiting process is carried by telephone, flyer, home page, personal meetings, and social media. The approach is convenience sampling.

Randomisation. In advance of the study, a randomisation concept determines the participant's random assignment to intervention or control group. The first half of the 220 participants are 70% likely to be assigned to the intervention group and 30% to the control group. For the second half of the sample the likelihood for group assignment reverses. This step should guarantee that enough participants receive the intervention in case of challenging recruitment. The intervention is favoured over an equal distribution to the groups. At the University Clinic of Neurology, where the examination takes place, only a study nurse knows about the group assignment of the patients, forwarding this information to the personnel of the SVDL and the ÖRK.

Blinding. In the context of the study, blinding of the employees of the SVDL and ÖRK is not possible since the intervention is apparent to the personnel. The neurologists and neuropsychologists are not informed at any time during the study of the patient's group assignment.

Intervention. "Multimodal Activation" (MMA) is an app developed for tablets that contains a serious game and has been previously tested in patients with dementia. It stimulates a multimodal training by games that involve cognitive and physical exercises. These exercises can be individually adapted to content, level of difficulty, sequence and time. The training starts with physical exercises accompanied by music. Afterwards there are cognitive exercises such as a quiz, puzzle, gap-filling, simple arithmetic tasks or listening comprehensions. The patients can use MMA at home as well as in a care facility.

Intervention group (IG). The IG undertakes a 1.5-year tablet PC-based training of cognitive and physical skills using DaheimAktiv, which is carried out every 14 days by a MAS trainer, medical nurse or pedagogically trained person from the SVDL or the ÖRK together with the patient. The tablet remains with the patient at home and the participants are encouraged to continue training without the presence of a trainer (with and without a relative). All training sessions are recorded. DaheimAktiv is a multimodal intervention procedure with cognitive and physical exercises. In addition to the fourteen-day training units with the trainers and independent training, "training cafés" will take place in small groups to promote motivation and increase social integration, i.e. several patients train together.

Control group (CG). In the control group, the medical interventions initiated are continued (standard intervention). Apart from that, these patients are subjected to the same study conditions as the patients of the intervention group. After completion of the evaluation phase, patients of the CG will receive a free, one-year license for DaheimAktiv.

Study outline. First, a pre-screening of potential participants takes place to check for inclusion and exclusion criteria. The patients that fit the criteria are invited to the University Clinic of Neurology for a neurological examination, blood sampling (also for potential genetic analysis) and cognitive assessments (performance tests and interviews). If a diagnosis of Alzheimer's disease is confirmed on a clinical basis, patients are invited to a structural and functional magnetic resonance imaging (MRI) in order to exclude other causes of cognitive deficits and aggregate imaging biomarkers of disease-associated changes such as hippocampal volume. Six and twelve months after study inclusion short cognitive testing and interviews at home will be carried out. After 1.5 years, the patients from the control and the intervention group again are invited to the University Clinic of Neurology performing the same procedures as during baseline.

Hotline. For the duration of the study, the SVDL provides a hotline specific for questions and problems that participants might face.

Statistics. The quantitative data will be analysed using IBM SPSS (version 25.0, 2017). The chosen level of significance is determined at α = .05. Mean and standard deviation or median and quartiles will be part of the descriptive statistics. Absolute and relative frequencies will depict categorical data. In order to test for the hypothesis regarding the positive effect of tablet training on cognition, primary outcome parameters (such as global neuropsychological scores) as well as secondary variables (such as neuropsychological subscores) will be compared between intervention and control group using ANCOVA adjusted for multiple testing. Furthermore, total brain volume, local volume of brain areas such as the hippocampus, cerebral microstructure and functional connectivity will be measured and compared between groups. Other secondary outcome parameters will be analysed using ANCOVA for between group comparisons. Pre-post comparisons (by ANOVA for repeated measures) shall deepen the understanding of how these changes occur over time. The analyses will be adjusted for age, sex, comorbidity and education. Qualitative data from the interviews will be organized and coded via the software MAXQDA. Afterwards a qualitative content analysis will be applied.

Ethics. Patients (or the person with power of attorney) have to give informed consent in order to participate in the study. At any given time, the participants can refuse or withdraw the consent without giving specific reasons. The genetic analysis merely serves a scientific purpose and requires written consent. All samples are analysed and stored using pseudonyms. Only at the University Clinic of Neurology it is possible to connect the sample with the name of the donor. If the results of the genetic analysis will be used for multi-centric research, it is ensured that the identity of the donor remains anonymous for cooperating centres. All aspects of the examination are non-invasive (except blood sampling), state-of-the-art procedures that are applied according to the law. The ethics committee of the Medical University of Graz approved the study on February 5th 2020 (31-556 ex 18/19).

Data protection Every participant receives an individual, pseudonymous code at the University Clinic of Neurology that is shared with the SVDL and ÖRK for patient-code assignment. The other partners of the study team only receive the patient's code. The communication between the project partners and all data transfer occurs using this code to ensure the anonymity of the patients. The SVDL submits questionnaires and interviews to the Medical University of Graz (MUG) via a secured server (protected by password). All personal information about the participants is confidential. Interviews are pseudonymised during transcription. The project partners have access to the data for the purpose of data entry and analysis.

For the tablet-based training with the MMA app, a registration with an email-address and a password is necessary. This information is stored in a coded form in a database. The serial number of the tablet has to be stored as well. Further personal information is optional and hence not required to use the training.

The app also stores information about every completed unit in the programme like speed and precision in the training intervention for the sake of future improvement. For further analysis of the intervention group, the data will be pseudonymous.

The usage of fitness trackers only works in combination with an account that the users have to create in the first place. However, there is no data transfer of the log data to the central database of the project. Only the users can access that data.

Trainings. In order to minimize the inter-rater variability of thr raters for questionnaires and interviews, the data-collecting persons of the SVDL and the ÖRK are trained beforehand on the questionnaires and interviews (individual interviews, focus groups) by employees of the MUG Neurology and nursing. For the tablet training, the SVDL and the ÖRK will train the dementia trainers to use the intervention. The duration will be about 4 hours. All participants/patients receive training in the application of the intervention by the SVDL/ÖRK.

Hotline, contact persons. During the study, the SVDL will set up a hotline for questions and problems of the participants during the study period. Regular times are given for this.

ELIGIBILITY:
Inclusion Criteria:

Persons with dementia

* are diagnosed of possible or probable dementia according to NINCDS-ADRDA criteria (McKhann et al. 2011).
* are older than 40 years at baseline examination.
* are able to speak and understand German and possesses sufficient physical, auditory and visual faculties to take part in a neuropsychological examination and a tablet-based training.
* have been receiving stable medication therapy for a minimum of 3 months before the baseline examination.
* who have been treated with a Memantine therapy, which started 3 months before the baseline examination.
* will be accompanied to the neurological examinations at T0a and T3a at the University Clinic of Neurology by an informal caregiver (relative or other significant person).
* may receive professional 24-hours-care - in this case an informal caregiver must be recruited as participant/accompanying person.
* live at home, with or without an informal caregiver (if alone, an informal caregiver should live nearby).
* receive professional care (e.g. home care services) or informal care (e.g. relatives) or no care yet.
* are willing and able to give informed consent or an informal caregiver with power of representation or a trustee gives the informed consent to participation in the study.
* do not receive any antipsychotic or antidepressive medication or have been stably adjusted to the medication for a minimum of 14 days before study start.

Informal caregivers

* are significant persons (e.g. family members, friends) of the participating persons with dementia (adults) which provide or do not provide care.
* living or not living with the person with dementia in the same household.
* are associated with a person with dementia receiving or not receiving professional care.
* speak and understand German.
* are able to give informed consent to participation in the study.

Dementia trainers

* are adults.
* are trained as M.A.S. (Morbus Alzheimer Syndrome) trainer.
* train the participants with dementia at home.
* speak and understand German.
* are able to give informed consent to participation in the study.

Exclusion Criteria

* Participation in a clinical trial until the last three months before study entry
* The participant presumably cannot finish the study
* Any of the following signs in brain MRI:

  * Infarct close to major vessels
  * More than one lacunar infarction (diameter 1.5cm in every spatial direction)
  * One lacunar infarct in a strategic region, such as the thalamus, the hippocampus or the caudate nucleus
  * Confluent lesions in deep white matter (Fazekas Score 3)
  * Other focal lesions potentially causing cognitive status (e.g. infections, lesions, normal pressure hydrocephalus)
* A general anesthetic three months before study entry or during study period
* The participant has a immunomodulating treatment or will receive a immunomodulating treatment during study period
* Cancer (last treatment >=5 years before study entry)
* Myocard infarction within 2 years before study entry
* Hepatitis B, C, HIV, Syphilis
* The patient has an active contagious disease
* The patient has a systemic disease potentially causing rapid progression

  * Insufficiently treated cardiac insufficiency (NYHA>3)
  * BMI>40
  * Insufficiently treated diabetes
  * Renal failure
  * Chronic liver disease
  * Other clinically relevant systemic diseases
* The Patient suffers from hypothyreosis. Patients with treated hypothyreosis may participate if stable therapy since >3 months is given
* Psychiatric diseases, such as schizophrenia, psychotic diseases or a bipolar disease

  * Current depressive episode or major depression within the last 2 years before study entry
* Metabolic or toxic encephalopathy or dementia due to general medical conditions

Ages: 50 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change of cognition (persons with dementia) | day 0, month 6, month 12, month 18
  The "Montreal Cognitive Assessment" has 30 items in 8 domains of cognitive functioning: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. 0-30 points can be obtained. Lower scores indicate a higher degree of cognitive impairment.
Neuropsychological Test Battery | day 0, month 18
  Pre-post comparisons in cognitive assessment's composite scores will used for efficacy of the tablet-training. The following z-transformed scores will be used to calculate a composite score:
  Wechsler Memory Scale (WMS-III-R) : Visuelle Paarerkennung I (min-ma:0-18, higher= better) Wechsler Memory Scale (WMS-III-R) : Verbale Paarerkennung I (min-ma:0-24, higher=better)
  Wechsler Memory Scale (WMS-III-R) : digit span (min-max:
  Trail Making Test, Version A (min-max: 0-180 seconds, lower better) Trail Making Test, Version B (min-max: 0-300 seconds, lower better) Verbaler Lern- und Merkfähigkeitstest, Subscore "Lernen und Datenakquisition" (min-ma:0-75, higher better) Testbatterie zur Aufmerksamkeitsprüfung (min-ma:0-n.a., lower better) Regensburger Wortflüssigkeitstest (verbal fluency test; 0-max, higher better); Letter Digit Subsitution Test (90 sec)
Change of cognition (persons with dementia) | day 0, month 6, month 12, month 18
  The Mini Mental Status Examination" (MMSE)

SECONDARY OUTCOMES:
Change of depression (persons with dementia) | day 0, month 18
  The short version of the "Geriatric Depression Scale" will be used for persons with dementia. The scale has 15 items (yes/no answers). 0-15 points can be obtained. Higher scores indicate a higher level of depressive symptoms.
Change of mobility (persons with dementia) | day 0, month 18
  The "Timed UP and GO Test" measures the time (in seconds) an individual needs to stand up from a standard arm chair, walk a distance of 3 meters, turn, walk back to the chair, and sit down. Interpretation: <10 seconds = completely unrestricted; 10-19 seconds = less mobile, but still unrestricted; 20 - 29 seconds = limited mobility; >30 seconds = pronounced mobility restriction. 14 seconds and more has been shown to indicate a high risk of falls.
Change of motivation (persons with dementia) | day 0, month 18 (AES self); day 0, month 6, month 12, month 18 (AES proxy, FAM)
  The "Apathy Evaluation Scale" is a scale to measure motivation because apathy can be understood as a loss of motivation. The scale has 18 items (4-point Likert scale). 18-72 points can be obtained. Higher scores correspond to a higher degree of apathy and therefore lower motivation. The German version (FAM) of the "Questionnaire on Current Motivation (QCM)" uses 18 items (7-point Likert scale) to measure the motivation to learn in terms of four motivational domains: anxiety, probability of success, interest, and challenge. The goal of the procedure is to prove the effects of current motivation on learning and performance. Four mean scale values are calculated. A total value is not calculated. For all subscales, higher levels on the respective subscales indicate a higher level of expression in the respective construct.
Change of quality of life (persons with dementia) | day 0, month 18
  The "Dementia Quality of Life Instrument" will be used for the participants with dementia. The instrument has 28 items (4-point Likert scale) and covers Quality of Life in the following three domains: emotions (items 1-13), memory (items 14-19) and activities of daily living (items 20-28). A global quality-of-life item is also included but does not contribute to the overall score. For every item, 1 to 4 points can be obtained, with higher scores indicating better quality of life.
Change of lifestyle factors (persons with dementia) | day 0, month 6, month 12, month 18
  The "Fantastic Lifestyle Checklist for Dementia (FANTASTIC-D)" is an instrument that assesses lifestyle factors of people with dementia. The instrument includes a total of 27 questions (5-point Likert scale) in the following 10 areas: 1) family, friends, 2) activity, 3) nutrition, 4) tobacco and toxins, 5) alcohol consumption, 6) sleep, shoes, stress 7) (type) personality 8) individual mental health 9) coping with role, situation 10) dementia-cognition. In total, between 0 and 108 points can be achieved with FANTASTIC-D. The higher the total score, the better the lifestyle of the respondent.
Technology acceptance (persons with dementia, informal caregivers, dementia trainers) | day 0, month 18; Interviews after 6 months
  The "Technology Usage Inventory" assesses participants' acceptance of new technologies and consists of 8 main domains: curiosity, anxiety, interest, user-friendliness, immersion, usefulness, skepticism, accessibility. These domains include 30 items using a 7-point Likert scale (ranging from 1=strongly disagree to 7=strongly agree). There is also a ninth domain "intention to use" with three items using a visual analogue scale: a straight horizontal line of 100 mm with the two ends (100 points=not agree; 0 points=agree). For all subscales, higher levels on the respective subscales indicate a higher level of expression in the respective construct. Individual interviews (people with dementia) and focus groups (other participants) will be conducted to obtain more in-deep knowledge.
Change of care dependency (persons with dementia) | day 0, month 18
  The "Care Dependency Scale" has 15 items (5-point Likert scale). 15-75 points can be obtained. Lower scores indicate a higher degree of care dependency.
Change of the activity level (persons with dementia) | day 0, month 18
  The "Pool Activity Level (PAL)" is a checklist to identify individuals' ability to engage in activity. It consists of nine everyday activities, with four activity levels: planned, exploratory, sensory and reflex. The description that most matches the individual's performance over the past two weeks is selected. The activity level that is most frequently ticked indicates the person's level of ability to engage in activity.
Change of care burden (informal caregivers) | day 0, month 18
  The "Zarid Burden Interview" captures the subjective burden of caregivers. The instrument has 22 items (5-point Likert scale). 0-88 points can be obtained. Higher scores indicate greater caregiver distress.
Change of perceived stress (informal caregivers) | day 0, month 18
  The Perceived Stress Scale (PSS-10) is a widely and well-established self-report scale measuring perceived stress. The PSS-10 measures the degree to which life in the past month has been experienced as unpredictable, uncontrollable and overwhelming on a 5-point Likert scale (0 = "never", 1="almost never", 2="sometimes", 3="fairly often", 4="very often"). Higher scores indicate a higher level of perceived stress.
Total Brain Volume measured with MRI | day 0, month 18
  Brain tissue volume, normalised for subject head size, will be estimated with SIENAX [Smith 2001, Smith 2002], part of FSL [Smith 2004]. SIENAX starts by extracting brain and skull images from the single whole-head input data [Smith 2002b]. The brain image is then affine-registered to MNI152 space [Jenkinson 2001, Jenkinson 2002] (using the skull image to determine the registration scaling); this is primarily in order to obtain the volumetric scaling factor, to be used as a normalisation for head size. Next, tissue-type segmentation with partial volume estimation is carried out [Zhang 2001] in order to calculate total volume of brain tissue (including separate estimates of volumes of grey matter, white matter, peripheral grey matter and ventricular CSF). Volume is then given as mm3.
Local Brain Volume measured with MRI | day 0, month 18
  FIRST is a model-based segmentation tool part of FSL [Smith 2004]. The shape models used in FIRST are constructed from manually segmented images provided by the Center for Morphometric Analysis (CMA), MGH, Boston. The manual labels are parameterized as surface meshes and modelled as a point distribution model. Deformable surfaces are used to automatically parameterize the volumetric labels in terms of meshes; the deformable surfaces are constrained to preserve vertex correspondence across the training data. Furthermore, normalized intensities along the surface normals are sampled and modelled. The shape and appearance model is based on multivariate Gaussian assumptions. Shape is then expressed as a mean with modes of variation (principal components). The investigators are primarily interested in the volume (mm3) of the hippocampus and the basal ganglia.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Koini, Principal Investigator — Medical University of Graz, Department of Neurology
Locations (1):
- Medical University of Graz, Austria, Graz, Styria, Austria

REFERENCES:
- [Background] Berwig M, Leicht H, Gertz HJ. Critical evaluation of self-rated quality of life in mild cognitive impairment and Alzheimer's disease--further evidence for the impact of anosognosia and global cognitive impairment. J Nutr Health Aging. 2009 Mar;13(3):226-30. doi: 10.1007/s12603-009-0063-4. PMID 19262958
- [Background] Berwig M, Leicht H, Hartwig K, Gertz HJ. Self-related quality of life in mild cognitive impairment and alzheimers disease. 2011; GeroPsych, 24(1):45-51.
- [Background] Braun M, Scholz U, Hornung R, Martin M. [Caregiver burden with dementia patients. A validation study of the German language version of the Zarit Burden Interview]. Z Gerontol Geriatr. 2010 Apr;43(2):111-9. doi: 10.1007/s00391-010-0097-6. Epub 2010 Mar 5. German. PMID 20204383
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Dijkstra A, Buist G, Dassen T. Nursing-care dependency. Development of an assessment scale for demented and mentally handicapped patients. Scand J Caring Sci. 1996;10(3):137-43. doi: 10.1111/j.1471-6712.1996.tb00326.x. PMID 9060783
- [Background] Gauggel S, Birkner B. Validität und Reliabilität einer deutschen Version der Geriatrischen Depressionsskala (GDS) [articel in German], Zeitschrift für Klinische Psychologie und Psychotherapie. 1999; 28:18-27.
- [Background] Klein EM, Brahler E, Dreier M, Reinecke L, Muller KW, Schmutzer G, Wolfling K, Beutel ME. The German version of the Perceived Stress Scale - psychometric characteristics in a representative German community sample. BMC Psychiatry. 2016 May 23;16:159. doi: 10.1186/s12888-016-0875-9. PMID 27216151
- [Background] Knorr C, Fröhlich L. What determines health related quality of life (HRQOL) in patients with dementia and their caregivers? International Society for Quality of Life Research meeting abstracts [http://www.isoqol.org/2007mtgabstracts.pdf]. Quality of Life Research supplement A-116, Abstract #1636 2007. 2007.
- [Background] Kothgassner OD, Felnhofer A, Hauk N, Kastenhofer E, Gomm J, Kryspin-Exner, I. TUI Technology Usage Inventory. ICARUS (Information- and Communication technology Applications: Research on User-oriented Solutions). 2013; Wien.
- [Background] Lohrmann C, Dijkstra A, Dassen T. Care dependency: testing the German version of the Care Dependency Scale in nursing homes and on geriatric wards. Scand J Caring Sci. 2003 Mar;17(1):51-6. doi: 10.1046/j.1471-6712.2003.00117.x. PMID 12581295
- [Background] Lueken U, Seidl U, Schwarz M, Volker L, Naumann D, Mattes K, Schroder J, Schweiger E. [Psychometric properties of a German version of the Apathy Evaluation Scale]. Fortschr Neurol Psychiatr. 2006 Dec;74(12):714-22. doi: 10.1055/s-2006-932164. German. PMID 17167730
- [Background] Marin RS, Biedrzycki RC, Firinciogullari S. Reliability and validity of the Apathy Evaluation Scale. Psychiatry Res. 1991 Aug;38(2):143-62. doi: 10.1016/0165-1781(91)90040-v. PMID 1754629
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Pool J. 2008. The pool activity level (PAL) instrument for occupational profiling : a practical resource for carers of people with cognitive impairment. London; Philadelphia: Jessica Kingsley Publishers.
- [Background] Rheinberg F, Vollmeyer R, Burns BD. FAM: Ein Fragebogen zur Erfassung aktueller Motivation in Lern- und Leistungssituationen. Diagnostica. 2001; 47(2):57-66.
- [Background] Smith SC, Lamping DL, Banerjee S, Harwood R, Foley B, Smith P, Cook JC, Murray J, Prince M, Levin E, Mann A, Knapp M. Measurement of health-related quality of life for people with dementia: development of a new instrument (DEMQOL) and an evaluation of current methodology. Health Technol Assess. 2005 Mar;9(10):1-93, iii-iv. doi: 10.3310/hta9100. PMID 15774233
- [Background] Tatzer VC, Pool J. Assessment: Pool Activity Level (PAL) - Aktivitätslevel bestimmen. Ergopraxis. 2018; 11(07/08):37-39
- [Background] Wilson DMC and Ciliska D, 1984. Lifestyle assessment: Development and use of the FANTASTIC checklist. Canadian Family Physician 30:1527-1532.
- [Background] Wilson DMC, Nielsen, E, Ciliska. Lifestyle Assessment: Testing the FANTASTIC Instrument. Can Fam Physican 1984; 30:1863-1866.
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Derived] Zuschnegg J, Ropele S, Opriessnig P, Schmidt R, Russegger S, Fellner M, Leitner M, Spat S, Garcia ML, Strobl B, Ploder K, Pszeida M, Hofmarcher-Holzhacker MM, Stoegerer-Oberschmid E, Guttmann-Lattmanig A, Paletta L, Schussler S, Koini M. The effect of tablet-based multimodal training on cognitive functioning in Alzheimer's disease: A randomized controlled trial. PLoS One. 2025 Aug 13;20(8):e0329931. doi: 10.1371/journal.pone.0329931. eCollection 2025. PMID 40802794